CLINICAL TRIAL: NCT00569946
Title: PHASE 2 STUDY OF AG-013736 AS SECOND-LINE TREATMENT IN PATIENTS WITH METASTATIC RENAL CELL CANCER
Brief Title: Study Of AG-013736 (Axitinib) As Second-Line Treatment In Patients With Metastatic Renal Cell Cancer (mRCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: A4061035
Record Dates: First submitted 2007-12-07; First posted 2007-12-10 (Estimated); Results first posted 2012-03-27 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-05

CONDITIONS: Carcinoma, Renal Cell
Keywords: AG-013736; RCC; Phase 2
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AG-013736 (Experimental)
  Interventions: Drug: AG-013736

INTERVENTIONS:
Drug: AG-013736 — AG-013736 5 mg BID will be administered orally on continuous schedule. Cycle length is 28 days. If the drug is well tolerated at 5 mg BID, the dose of AG-013736 may be titrated to 7 mg BID and then to a maximum of 10 mg BID.
  Number of cycles: until progression or unacceptable toxicity develops.

SUMMARY:
To investigate objective tumor response of AG-013736 for metastatic Renal Cell Cancer (mRCC)

ELIGIBILITY:
Inclusion Criteria:

* Patients histologically diagnosed as metastatic renal cell cancer with a component of clear cell cancer.
* Patients who are refractory to cytokine therapy as 1st line.
* Patients who experienced nephrectomy.
* Patients with at least 1 target lesion, as defined by RECIST.
* Patients with no uncontrolled hypertension.

Exclusion Criteria:

* Gastrointestinal abnormalities
* Current use or anticipated inability to avoid potent CYP3A4 inhibitors or CYP1A2/3A4 inducers.
* Active seizure disorder or evidence of brain metastases.
* Patients with hemoptysis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-12-12 (Actual); Primary Completion 2010-02-26 (Actual); Study Completion 2012-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- Japan (18):
  - National Cancer Center East Hospital, Kashiwa, Chiba
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Tsukuba University Hospital, Tsukuba, Ibaraki
  - Iwate Medical University, Morioka, Iwate
  - Kochi Medical School Hospital, Nankoku-shi, Kochi
  - Kinki University Hospital, Sayama, Osaka
  - Hamamatsu University School of Medicine University Hospital, Hamamatsu, Shizuoka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Tokyo Women's Medical University Medical Center East, Arakawa-ku, Tokyo
  - National Cancer Center, Chuo-ku, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - Akita University Hospital, Akita
  - National Kyushu Cancer Center, Fukuoka
  - Kyushu University Hospital, Department of Urology, Fukuoka
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Osaka University Hospital, Osaka
  - Tokushima University Hospotal, Tokushima
  - Yamagata University Hospital, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Schindler E, Amantea MA, Karlsson MO, Friberg LE. A Pharmacometric Framework for Axitinib Exposure, Efficacy, and Safety in Metastatic Renal Cell Carcinoma Patients. CPT Pharmacometrics Syst Pharmacol. 2017 Jun;6(6):373-382. doi: 10.1002/psp4.12193. Epub 2017 May 26. PMID 28378918
- [Derived] Eto M, Uemura H, Tomita Y, Kanayama H, Shinohara N, Kamei Y, Fujii Y, Umeyama Y, Ozono S, Naito S, Akaza H; Japan Axitinib Phase II Study Group. Overall survival and final efficacy and safety results from a Japanese phase II study of axitinib in cytokine-refractory metastatic renal cell carcinoma. Cancer Sci. 2014 Dec;105(12):1576-83. doi: 10.1111/cas.12546. Epub 2014 Nov 25. PMID 25283266
- [Derived] Tomita Y, Uemura H, Fujimoto H, Kanayama HO, Shinohara N, Nakazawa H, Imai K, Umeyama Y, Ozono S, Naito S, Akaza H; Japan Axitinib Phase II Study Group. Key predictive factors of axitinib (AG-013736)-induced proteinuria and efficacy: a phase II study in Japanese patients with cytokine-refractory metastatic renal cell Carcinoma. Eur J Cancer. 2011 Nov;47(17):2592-602. doi: 10.1016/j.ejca.2011.07.014. Epub 2011 Aug 31. PMID 21889330
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061035&StudyName=Study%20Of%20AG-013736%20%28Axitinib%29%20As%20Second-Line%20Treatment%20In%20Patients%20With%20Metastatic%20Renal%20Cell%20Cancer%20%28mRCC%29%0A

RESULTS

PARTICIPANT FLOW:
Groups:
- AG-013736: The starting dose of AG-013736 was 5 mg twice daily (BID), which was administered orally at approximately 12 hours apart in cycles of 4 weeks (28 days). The treatment is to be continued until the participants meet the discontinuation criteria such as disease progression or intolerable toxicity. The dose of AG-013736 could be titrated to 7 mg BID, and then 10 mg BID or reduced to 3 mg BID, and then 2 mg BID depending on the grade, type, and causality of adverse events experienced.
Period: Overall Study
Arm/Group | AG-013736
Started | 64
Completed | 5
Not Completed | 59
Not completed — Adverse Event | 16
Not completed — Objective Progression or Relapse | 42
Not completed — Global Deterioration of Health Status | 1

BASELINE CHARACTERISTICS:
Arm/Group | AG-013736
Number analyzed (Participants) | 64
Age, Customized [Count of Participants; unit: Participants]
  <18 | 0
  18-44 | 6
  45-64 | 30
  >= 65 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 44

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (Percentage of Participants With Complete Response [CR] or Partial Response [PR]): Independent Review Committee Assessment
Description: Percentage of participants with objective response based assessment of confirmed CR or confirmed PR by the Independent Review Committee, according to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.0). CR was defined as the disappearance of all target and nontarget lesions and no appearance of new lesions. PR was defined as at least a 30% decrease in the sum of the longest diameters of the targeted lesions. CR and PR had to be documented on 2 occasions separated by at least 4 weeks.
Time Frame: Up to 765 days of treatment at the data cut-off date
Population: The Intent-To-Treat (ITT) population included all participants enrolled in the study who received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AG-013736
Number analyzed (Participants) | 64
percentage of participants | 50.0 [37.2 to 62.8]

2. Primary Outcome: Objective Response Rate (Percentage of Participants With Complete Response [CR] or Partial Response [PR]): Investigators Assessment
Description: Percentage of participants with objective response based assessment of confirmed CR or confirmed PR by the investigator, according to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.0). CR was defined as the disappearance of all target and nontarget lesions and no appearance of new lesions. PR was defined as at least a 30% decrease in the sum of the longest diameters of the targeted lesions. CR and PR had to be documented on 2 occasions separated by at least 4 weeks.
Time Frame: Up to 765 days of treatment at the data cut-off date
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AG-013736
Number analyzed (Participants) | 64
percentage of participants | 54.7 [41.7 to 67.2]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: Time in months from start of study treatment to first documentation of objective tumor progression or death due to any cause whichever comes first. PFS was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 30.44. Tumor progression was determined from radiological image (where data meet the criteria for progressive disease [PD]).
Time Frame: Up to 1709 days of treatment
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AG-013736
Number analyzed (Participants) | 64
months
  Independent Review Committee Assessment | 11.0 [9.2 to 12.0]
  Investigators Assessment | 12.0 [9.2 to 14.8]

4. Secondary Outcome: Time to Tumor Progression (TTP)
Description: Time in months from start of study treatment to first documentation of objective tumor progression. TTP was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 30.44. Tumor progression was determined from radiological image (where data meet the criteria for progressive disease [PD]).
Time Frame: Up to 1709 days of treatment
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AG-013736
Number analyzed (Participants) | 64
months
  Independent Review Committee Assessment | 11.0 [9.2 to 12.0]
  Investigators Assessment | 12.0 [9.2 to 14.8]

5. Secondary Outcome: Duration of Response
Description: Time in months from the first documentation of objective tumor response to objective tumor progression or death due to any cause. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 30.44. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: Start of first confirmed CR or PR to the date of the first event (PD or death) or the last tumor assessment, whichever came first, assessed up to 1709 days.
Population: The Intent-To-Treat (ITT) population included all participants enrolled in the study who received at least 1 dose of study medication. DR was calculated for the subgroup of participants with a confirmed objective tumor response. n=number of participants assessed as CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AG-013736
Number analyzed (Participants) | 64
months
  Independent Review Committee Assessment (n=33) | 11.1 [8.2 to 13.7]
  Investigators Assessment (n=36) | 12.8 [7.7 to 17.5]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of first dose of AG-013736 to date of death due to any cause.
  Subjects in whom death is not reported will have their event time censored on the last date the subject is known to be alive.
Time Frame: Up to 2002 days (maximum duration of treatment plus follow-up observation)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AG-013736
Number analyzed (Participants) | 64
months | 37.3 [28.6 to 49.9]

7. Secondary Outcome: Number of Participants Analyzed for Population Pharmacokinetics of AG-013736
Description: Population pharmacokinetic analysis of AG-013736 is conducted by combining current study data with other AG-013736 studies.
Time Frame: Cycle 1 Day 1 (2 hours after morning dose); Cycles 3, 5, and 7 Day 1 predose and 2 hours post morning dose
Population: No population pharmacokinetic analysis results are available just for the current study.
Arm/Group | AG-013736
Number analyzed (Participants) | 0

8. Secondary Outcome: Plasma Concentration of Soluble Vascular Endothelial Growth Factor Receptor 1 (s-VEGFR1)
Time Frame: Cycle 1 Day 1 predose, Day 1 of Cycle 2 to Cycle 7, and end of treatment/discontinuation (assessed up to 1709 days)
Population: Biomarker analysis set included all participants enrolled in the study who received at least 1 dose of study medication and who submitted at least 1 sample; n=number of participants assessed.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | AG-013736
Number analyzed (Participants) | 64
pg/mL
  Cycle 1 Day 1 (n=64) | 83.10 [44.3 to 215]
  Cycle 2 Day 1 (n=63) | 63.60 [0 to 190]
  Cycle 3 Day 1 (n=60) | 68.20 [36.4 to 936]
  Cycle 4 Day 1 (n=59) | 69.20 [33.5 to 119]
  Cycle 5 Day 1 (n=57) | 62.90 [0 to 125]
  Cycle 6 Day 1 (n=52) | 62.00 [32.1 to 119]
  Cycle 7 Day 1 (n=48) | 57.75 [0 to 101]
  End of Treatment/Discontinuation (n=55) | 76.60 [0 to 2780]

9. Secondary Outcome: Plasma Concentration of Soluble Vascular Endothelial Growth Factor Receptor 2 (s-VEGFR2)
Time Frame: Cycle 1 Day 1 predose, Day 1 of Cycle 2 to Cycle 7, and end of treatment/discontinuation (assessed up to 1709 days)
Population: as for outcome 8
Measure: Median (Full Range); unit: pg/mL
Arm/Group | AG-013736
Number analyzed (Participants) | 64
pg/mL
  Cycle 1 Day 1 (n=64) | 8900.0 [2620 to 13400]
  Cycle 2 Day 1 (n=63) | 6040.0 [2760 to 12600]
  Cycle 3 Day 1 (n=60) | 5980.0 [3340 to 11600]
  Cycle 4 Day 1 (n=59) | 6030.0 [3310 to 11600]
  Cycle 5 Day 1 (n=57) | 5880.0 [3140 to 10400]
  Cycle 6 Day 1 (n=52) | 5790.0 [3160 to 9920]
  Cycle 7 Day 1 (n=48) | 5395.0 [3620 to 10400]
  End of Treatment/Discontinuation (n=55) | 6540.0 [2870 to 12600]

10. Secondary Outcome: Plasma Concentration of Soluble Vascular Endothelial Growth Factor Receptor 3 (s-VEGFR3)
Time Frame: Cycle 1 Day 1 predose, Day 1 of Cycle 2 to Cycle 7, and end of treatment/discontinuation (assessed up to 1709 days)
Population: as for outcome 8
Measure: Median (Full Range); unit: pg/mL
Arm/Group | AG-013736
Number analyzed (Participants) | 64
pg/mL
  Cycle 1 Day 1 (n=64) | 20250.0 [2060 to 132000]
  Cycle 2 Day 1 (n=63) | 12000.0 [1990 to 45700]
  Cycle 3 Day 1 (n=60) | 13100.0 [2090 to 47700]
  Cycle 4 Day 1 (n=59) | 13800.0 [0 to 39100]
  Cycle 5 Day 1 (n=57) | 16700.0 [0 to 38100]
  Cycle 6 Day 1 (n=52) | 15550.0 [5200 to 39800]
  Cycle 7 Day 1 (n=48) | 13750.0 [0 to 38200]
  End of Treatment/Discontinuation (n=55) | 22300.0 [0 to 54500]

11. Secondary Outcome: Plasma Concentration of Soluble Stem Cell Factor Receptor (s-KIT)
Time Frame: Cycle 1 Day 1 predose, Day 1 of Cycle 2 to Cycle 7, and end of treatment/discontinuation (assessed up to 1709 days)
Population: as for outcome 8
Measure: Median (Full Range); unit: pg/mL
Arm/Group | AG-013736
Number analyzed (Participants) | 64
pg/mL
  Cycle 1 Day 1 (n=64) | 39050.0 [24800 to 73700]
  Cycle 2 Day 1 (n=63) | 35000.0 [21800 to 64000]
  Cycle 3 Day 1 (n=60) | 37300.0 [20700 to 65000]
  Cycle 4 Day 1 (n=59) | 38100.0 [20100 to 64300]
  Cycle 5 Day 1 (n=57) | 39800.0 [24600 to 70700]
  Cycle 6 Day 1 (n=52) | 41400.0 [23500 to 65900]
  Cycle 7 Day 1 (n=48) | 42400.0 [23100 to 62000]
  End of Treatment/Discontinuation (n=55) | 40600.0 [22200 to 72000]

12. Secondary Outcome: Plasma Concentration of Vascular Endothelial Growth Factor (VEGF)
Time Frame: Cycle 1 Day 1 predose, Day 1 of Cycle 2 to Cycle 7, and end of treatment/discontinuation (assessed up to 1709 days)
Population: as for outcome 8
Measure: Median (Full Range); unit: pg/mL
Arm/Group | AG-013736
Number analyzed (Participants) | 64
pg/mL
  Cycle 1 Day 1 (n=64) | 63.40 [26.4 to 361]
  Cycle 2 Day 1 (n=63) | 162.00 [31.5 to 856]
  Cycle 3 Day 1 (n=60) | 137.00 [26.3 to 723]
  Cycle 4 Day 1 (n=59) | 145.00 [21.9 to 514]
  Cycle 5 Day 1 (n=57) | 155.00 [24.3 to 554]
  Cycle 6 Day 1 (n=52) | 184.50 [21.3 to 743]
  Cycle 7 Day 1 (n=48) | 180.00 [46 to 762]
  End of Treatment/Discontinuation (n=55) | 121.00 [15.6 to 617]

13. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with any adverse events, adverse events graded as Common Terminology Criteria (CTCAE) for Adverse Events Version 3.0 Grade 3 or higher , serious adverse events, or adverse events resulted in discontinuation.
Time Frame: Up to 1709 days of treatment plus 28-days follow-up
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | AG-013736
Number analyzed (Participants) | 64
participants
  Any adverse events | 64
  Any serious adverse events | 21
  Any Grade-3 or -4 adverse events | 58
  Any Grade-5 adverse events (= death) | 1
  Discontinuation due to adverse events | 16

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | AG-013736
Serious Adverse Events (participants affected / at risk) | 21/64
Other Adverse Events (participants affected / at risk) | 64/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AG-013736 (N=64)
Acute myocardial infarction (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Duodenal stenosis (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Peptic ulcer (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Disease progression (General disorders) | 1
Malaise (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Appendicitis (Infections and infestations) | 1
Cryptococcosis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pyelonephritis (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Balance disorder (Nervous system disorders) | 1
Leukoencephalopathy (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AG-013736 (N=64)
Anaemia (Blood and lymphatic system disorders) | 5
Leukocytosis (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Polycythaemia (Blood and lymphatic system disorders) | 3
Angina pectoris (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 2
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 3
Ear haemorrhage (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 3
External ear pain (Ear and labyrinth disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Otorrhoea (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 5
Vertigo (Ear and labyrinth disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 2
Hypothyroidism (Endocrine disorders) | 31
Blepharitis (Eye disorders) | 1
Cataract (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Conjunctivitis allergic (Eye disorders) | 1
Dry eye (Eye disorders) | 2
Eye discharge (Eye disorders) | 2
Eye pain (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 2
Eyelid pain (Eye disorders) | 1
Pinguecula (Eye disorders) | 1
Retinal haemorrhage (Eye disorders) | 1
Retinal tear (Eye disorders) | 1
Retinal vein occlusion (Eye disorders) | 1
Vision blurred (Eye disorders) | 2
Visual acuity reduced (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 9
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 9
Anal fistula (Gastrointestinal disorders) | 1
Anal pruritus (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 14
Dental caries (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 44
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 3
Duodenal ulcer (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 5
Epigastric discomfort (Gastrointestinal disorders) | 1
Faecal incontinence (Gastrointestinal disorders) | 1
Gastric polyps (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 6
Gingival bleeding (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Gingival swelling (Gastrointestinal disorders) | 1
Glossitis (Gastrointestinal disorders) | 2
Glossodynia (Gastrointestinal disorders) | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 4
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 22
Oral pain (Gastrointestinal disorders) | 2
Paraesthesia oral (Gastrointestinal disorders) | 3
Perianal erythema (Gastrointestinal disorders) | 1
Periodontal disease (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 15
Tongue disorder (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 12
Chest discomfort (General disorders) | 3
Chest pain (General disorders) | 10
Chills (General disorders) | 2
Disease progression (General disorders) | 1
Face oedema (General disorders) | 4
Fatigue (General disorders) | 36
Gait disturbance (General disorders) | 1
Hypothermia (General disorders) | 2
Influenza like illness (General disorders) | 3
Local swelling (General disorders) | 1
Malaise (General disorders) | 9
Medical device complication (General disorders) | 1
Mucosal inflammation (General disorders) | 4
Oedema (General disorders) | 6
Oedema peripheral (General disorders) | 7
Pain (General disorders) | 2
Puncture site pain (General disorders) | 1
Pyrexia (General disorders) | 10
Thirst (General disorders) | 1
Ulcer (General disorders) | 1
Alcoholic liver disease (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 8
Hyperbilirubinaemia (Hepatobiliary disorders) | 3
Liver disorder (Hepatobiliary disorders) | 1
Contrast media allergy (Immune system disorders) | 1
Acute sinusitis (Infections and infestations) | 1
Adenoiditis (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Cystitis (Infections and infestations) | 4
Folliculitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 4
Gastroenteritis viral (Infections and infestations) | 2
Genital infection fungal (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 4
Herpes zoster (Infections and infestations) | 4
Hordeolum (Infections and infestations) | 3
Infected dermal cyst (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 25
Onychomycosis (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 9
Pharyngitis (Infections and infestations) | 1
Pulpitis dental (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 3
Skin candida (Infections and infestations) | 2
Tinea infection (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 6
Laceration (Injury, poisoning and procedural complications) | 1
Ligament injury (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Scratch (Injury, poisoning and procedural complications) | 1
Tooth injury (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Wound complication (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 15
Amylase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 15
Blood albumin decreased (Investigations) | 7
Blood alkaline phosphatase increased (Investigations) | 13
Blood calcium decreased (Investigations) | 2
Blood chloride decreased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 5
Blood lactate dehydrogenase increased (Investigations) | 8
Blood potassium increased (Investigations) | 2
Blood pressure decreased (Investigations) | 1
Blood sodium decreased (Investigations) | 2
Blood thyroid stimulating hormone decreased (Investigations) | 4
Blood thyroid stimulating hormone increased (Investigations) | 21
Blood urea decreased (Investigations) | 1
Blood urea increased (Investigations) | 6
Blood uric acid increased (Investigations) | 1
Blood urine present (Investigations) | 5
C-reactive protein increased (Investigations) | 7
Gamma-glutamyltransferase increased (Investigations) | 3
Haematocrit decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 5
International normalised ratio increased (Investigations) | 2
Liver function test abnormal (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 8
Protein total decreased (Investigations) | 1
Protein urine (Investigations) | 5
Protein urine present (Investigations) | 2
Prothrombin time shortened (Investigations) | 1
Red blood cell count decreased (Investigations) | 2
Red blood cell count increased (Investigations) | 1
Thyroxine free decreased (Investigations) | 3
Thyroxine free increased (Investigations) | 3
Tri-iodothyronine free decreased (Investigations) | 1
Tri-iodothyronine free increased (Investigations) | 3
Weight decreased (Investigations) | 21
White blood cell count decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 27
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 15
Back pain (Musculoskeletal and connective tissue disorders) | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Altered state of consciousness (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 7
Dysgeusia (Nervous system disorders) | 12
Epilepsy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 18
Hyperaesthesia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 5
Neuropathy peripheral (Nervous system disorders) | 1
Parosmia (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 4
Mood altered (Psychiatric disorders) | 1
Panic disorder with agoraphobia (Psychiatric disorders) | 1
Bladder irritation (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 33
Renal impairment (Renal and urinary disorders) | 2
Genital tract inflammation (Reproductive system and breast disorders) | 1
Menstruation irregular (Reproductive system and breast disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 1
Scrotal haematocoele (Reproductive system and breast disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 34
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 3
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4
Acne (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 5
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Eczema (Skin and subcutaneous tissue disorders) | 3
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 2
Hair disorder (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 48
Penile ulceration (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 17
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Skin mass (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 56
Hypotension (Vascular disorders) | 1
Pneumonia (Infections and infestations) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Dysuria (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.